CLINICAL TRIAL: NCT07313657
Title: Integrating Mental Health Into Heart Failure Care: A Hybrid Type 1 Pretest-Posttest Feasibility Study of the FRAME Intervention
Brief Title: Improving Care and Mental Well-Being for Adults With Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: M16-25-028
Record Dates: First submitted 2025-09-23; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Mental Health; Stress; Anxiety; Depression
Keywords: Heart Failure and Mental Health
MeSH Terms: conditions — Heart Failure; Psychological Well-Being; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Hybrid Type 1 effectiveness- implementation design, which is well-suited to for evaluating interventions in real-world healthcare settings where both clinical outcomes and implementation processes are focus areas. This design evaluates the effectiveness of an intervention while also collecting formative data to understand it's implementation context, where we determine its feasibility, acceptability, barriers and facilitators to uptake to support future trials. The primary aim of Hybrid Type 1 would be to determine whether an intervention is effective in improving targeted outcomes. In our study, the aim of this design would be to determine whether the intervention is effective in improving our outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FRAME Intervention (Other): Every participant who completed the intake survey for baseline data collection will receive the FRAME intervention via email in January 2026.
  Interventions: Other: Heart Failure and Mental Health Intervention (FRAME)

INTERVENTIONS:
Other: Heart Failure and Mental Health Intervention (FRAME) — Foundation, Recognition, Awareness, Management and Engagement (FRAME) is a multi-component, co-designed web tool created in collaboration with patient partners, caregivers, healthcare providers, and Archipel and Great River Ontario Health Teams. It is designed to improve recognition, awareness, management and support for mental health in patients with heart failure. There are three different versions: one for healthcare providers, one for caregivers and one for patients. The intervention includes educational material about heart failure and mental health, conversational support to help facilitate discussions about mental health, self-management activity maps (e.g., tips about nutrition and exercise), asset maps (i.e., displaying available resources), and the provider-facing discussion tool to help initiate conversations about mental health and guide referrals or supports. FRAME was developed through a co-design process informed by the lived experiences of community partners.

SUMMARY:
Heart failure is a high-risk, chronic condition that impacts patients' mental health. Approximately 50% of heart failure patients experience comorbid mental health conditions, such as stress, depression and anxiety, which affect their day-to-day lives. Despite this interconnection, the integration of mental health awareness and support into cardiac care remains limited. To address this gap, the FRAME (Foundation, Recognition, Awareness, Management, Engagement) intervention was co-designed by researchers, healthcare providers, health system decisionmakers, and patient partners. This pilot study evaluates the feasibility of implementing the FRAME intervention in pilot clinical sites within two health regions in Ontario, Canada, including team-based family medicine clinics, cardiac rehabilitation/specialist clinics, and emergency departments. Utilizing a pretest-posttest hybrid 1 model intervention design, this study evaluates process indicators and patient-focused outcomes through surveys and semi-structured qualitative interviews. Findings from this study will inform a future large scale cohort study and scalable integration of the FRAME tool into existing cardiac care pathways to enhance mental health awareness and support among heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

For Patients (Surveys and Optional Interviews):

* Patients at risk of heart failure (e.g., irregular heartbeat, coronary artery disease, a past heart attack, high blood pressure that is being treated, cardiomyopathy), or with a self-reported/documented diagnosis of heart failure OR on the following list of medications :

  * Angiotensin receptor-neprilysin inhibitors (ARNI), called sacubitril-valsartan
  * Angiotensin converting enzyme inhibitors (ACEi), called "prils"
  * Angiotensin-receptor blockers (ARBs), called "sartans"
  * Beta-blockers, called "lols"
  * Mineralocorticoid receptor antagonists (MRAs)
  * Sodium-glucose co-transporter-2 (SGLT2) inhibitors, called "flozins"
* Receiving care at one of the participating pilot test sites or if they found their way to the tool website
* Willing and able to provide informed consent and name, email address and phone number for follow-up contact (for survey and interview)

Caregivers (Optional interviews):

* Caregivers who support adult(s) with heart failure.

Exclusion Criteria:

* Inability to provide informed consent (e.g., due to cognitive impairment or language barriers without translated support)
* Participants who do not have access to the internet will not be able to use the web-tool.

For Healthcare Providers

* Providers that are not involved in the care of heart failure patients

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7300 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of Mental Health Conversations | Baseline, and up to 6 months following intervention
  This outcome measures whether patients with heart failure report having a discussion about mental health with their healthcare provider or loved ones after being introduced to FRAME. This will be measured by changes in response to two questions in a survey given to participants pre- and post-intervention. These questions will ask if in the past 6 months, they have discussed mental health with a healthcare provider or if in the past 6 months, they have discussed mental health with their loved ones. The responses will include strongly disagree, disagree, neutral, agree and strongly agree. The intervention will be rolled out, after which they can respond to the post-intervention survey anytime until the study closes. Change in response from pre-intervention to post-intervention will be assessed.

SECONDARY OUTCOMES:
Engagement in Health Seeking Behaviours | Baseline, and up to 6 months following intervention
  This outcome evaluates whether participants (patients) report accessing mental health-related support, following the FRAME intervention. Supports may include formal resources (e.g., referrals to psychological services), informal or community-based support (e.g., peer groups, faith-based programs), and self-management strategies (e.g., mindfulness, exercise, online tools). This outcome will be measured in pre-post intervention surveys with the participants. The question will ask if, in the past 6 months, they have used community-based supports or if, in the past 6 months, they have used self-management strategies. Below these questions, there will be a list of the supports/strategies, and beside them will be checkboxes with the frequency of access. The options for this will be N/A, never, once, 2-3 times, every month and weekly or more. Change in response from pre-intervention to post-intervention will be assessed.
Confidence in Engaging in Mental Health Conversations and Knowledge of Mental Health | Baseline, and up to 6 months following intervention
  This outcome assesses perceived knowledge of the interconnection between mental health and heart failure through self-reported confidence in initiating mental health discussions. This outcome will be assessed through pre- and post-intervention surveys. The question assessing perceived knowledge of mental health will be about whether they know where to find information/support about mental health in their community. The question assessing confidence in engaging in mental health conversations will ask if they feel confident bringing up my mental health with a healthcare provider in a medical setting. Both questions will have checkbox options from strongly disagree to strongly agree, where a change in responses will be assessed from pre-intervention to post-intervention.

CONTACTS AND LOCATIONS:
Locations (9):
- Canada (9):
  - Seaway Valley Community Health Centre (Cardiac Rehab Program), Cornwall, Ontario
  - Centre de Santé Communautaire de l'Estrie, Limoges, Ontario
  - Orleans Cardiopulmonary Clinic, Orléans, Ontario
  - Bruyère Health Research Institute, Ottawa, Ontario
  - Byward Family Health Team, Ottawa, Ontario
  - Montfort Hospital, and associated Aline-Chrétien Rehabilitation Clinic, Ottawa, Ontario
  - Ste-Anne Medical Clinic, Ottawa, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Winchester Memorial Hospital, Winchester, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
We currently have no motivation for sharing IPD, but if our data becomes helpful for the conduction of a follow-up project, IPD may be shared.

REFERENCES:
- See also: Project Background and Information from the Research Team conducting this study — https://www.ccaeresearch.ca/brain-heart-interconnectome/
- See also: Project Background and Information from the Brain-Heart Interconnectome at the University of Ottawa — https://www.uottawa.ca/research-innovation/bhi/research/theme-4-innovative-health-systems-tailored-models-care

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT07313657/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT07313657/ICF_001.pdf